CLINICAL TRIAL: NCT06979258
Title: Heat Stress: Exposure Among Low-Income Residents in Bangladesh and Evaluation of Indoor Interventions
Brief Title: Heat Stress Exposure Among Low-Income Residents in Bangladesh and Evaluation of Indoor Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-08-17719; 1R01ES035910 (NIH)
Record Dates: First submitted 2025-04-25; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Heat Stress
Keywords: heat stress; cooling; heart rate; heart rate variability; sleep quality; Bangladesh
MeSH Terms: conditions — Heat Stress Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indoor cooling intervention (Experimental): Households in this arm will receive infrastructure and/or equipment intended to cool the house in the hot season.
  Interventions: Other: Cooling intervention
- Control (No Intervention): Households in this arm will not receive any intervention

INTERVENTIONS:
Other: Cooling intervention — Infrastructure and/or equipment that cools the house in the hot season
  Arms: Indoor cooling intervention

SUMMARY:
The goal of this clinical trial is to learn if infrastructure and equipment installed to cool homes reduce adverse health outcomes. The main questions it aims to answer are:

What is the impact of the intervention on indoor heat stress? What is the impact of the intervention on personal exposure to heat stress? What is the impact of the intervention on health outcomes, including heart rate, and heart rate variability, and sleep quality?

Participants will have cooling infrastructure and/or equipment installed in their home; have heat stress sensors installed inside and outside their home and wear personal heat stress monitors; allow some biological functions such as heat rate, heat rate variability, and sleep quality.

DETAILED DESCRIPTION:
During the last two decades, nearly half a million people died each year from heat-related causes; climate change is expected to exacerbate the burden of adverse health outcomes. Heat stress has been associated with an increase in all-cause mortality, cardiovascular disease and mortality, chronic respiratory disease, lower respiratory infection, chronic kidney disease, diabetes, adverse pregnancy outcomes, and poor mental health. The investigators will to determine personal heat stress of low-income individuals who do not have access to air conditioning, evaluate the effectiveness, acceptability, feasibility, and scalability of building-level cooling strategies to reduce indoor heat stress among vulnerable individuals, and evaluate the impact of these interventions on heart rate. A disproportionate burden of heat-related death and disease is borne by low-income communities because they do not have access to cooling and suffer from comorbidities that exacerbate the adverse impacts of heat stress. South Asia faces the greatest current and predicted loss in disability-adjusted life years due to heat stress, and heat stress is particularly strong in informal settlements. As such, the investigators plan to conduct this study in informal settlements in Dhaka, Bangladesh. The overall hypothesis is that individuals who live in homes with corrugated iron roofs and walls are at elevated risk of heat stress and that it is possible to modify homes to prevent increases in heart rate associated with heat stress, ultimately reducing cardiovascular morbidity and mortality. The investigators will evaluate the impact of cooling infrastructure and/or equipment interventions on residents' heart rate (primary outcome), heart rate variability, sleep quality, self-reported thermal comfort, mental health, wellness, fatigue, and indoor thermal conditions (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria for the house:

* House is located in an informal settlement in an urban area in Bangladesh
* The house has a corrugated iron roof and corrugated iron walls
* The household plans to remain in the house from Feb-Nov

Exclusion Criteria for the house

* There is an inhabited structure about the house
* The landlord does not allow the proposed intervention

Inclusion Criteria for the participant:

* Lives in an eligible household

Exclusion Criteria for the participant

* Has access to air conditioning in their home or place of work
* Reports they are pregnant
* Has hypertension, as measured by study staff
* Has diabetes, as measured by study staff
* Self-reports cardiovascular disease / chronic cardiac condition
* Self-reports respiratory disease / chronic respiratory condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1539 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 0, 2, and 4 weeks
  resting heart rate (beats per minute, bpm), where lower heart rate is better

SECONDARY OUTCOMES:
Heart rate variability | 0, 2, and 4 weeks
  resting heart rate (beats per minute, bpm) variability, where higher variability is better
Sleep quality | 0, 2, and 4 weeks
  Self-reported sleep quality and number of minutes in rapid eye movement (REM), as recorded by a fitness watch, where more time in REM is better
Irritability | 0, 2, and 4 weeks
  Self-reported irritability, as measured by the Brief Irritability Test (BITe), where a lower score is better
Environmental Symptoms | 0, 2, and 4 weeks
  Environmental symptoms, as measured by the abbreviated environmental symptoms questionnaire, where a lower score is better
Depression | 0, 2, and 4 weeks
  Depression as measured by the Patient Health Questionnaire version with 8 questions (PHQ-8). A total PHQ-8 score of >=7 indicated depression, >= 10 indicates major depression and >= 20 indicates severe depression.
Anxiety | 0, 2, and 4 weeks
  Anxiety, as measured by the Generalised Anxiety Disorder with 7 questions (GAD-7). A total GAD-7 score of >= 8 indicates anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Laura H Kwong, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be stored in icddrb's data repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The investigators expect the data to become available at least by 1 Jan 2030. The investigators have no plan for when the data will become unavailable.
Access Criteria: Reasonable request